CLINICAL TRIAL: NCT04284553
Title: Optimizing Electronic Health Record Prompts With Behavioral Economics to Improve Prescribing for Older Adults
Acronym: NUDGE-EHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Atrius Health (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Niteesh K. Choudhry, MD, PhD, Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019P002167
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Aging; Benzodiazepine Sedative Adverse Reaction; Anticholinergic Adverse Reaction; Adverse Drug Event
Keywords: Benzodiazepine; Sedative hypnotic; Overprescribing; Anticholinergic
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Medical Order Entry Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Base Order Entry Alert (Experimental)
  Interventions: Other: Order Entry; Other: Enhanced Alert
- Base Open Encounter Alert (Experimental)
  Interventions: Other: Open Encounter; Other: Enhanced Alert
- Order Entry + Follow-up booster Alert (Experimental)
  Interventions: Other: Order Entry; Other: Follow-up booster Alert; Other: Enhanced Alert
- Open Encounter + Follow-up booster Alert (Experimental)
  Interventions: Other: Open Encounter; Other: Follow-up booster Alert; Other: Enhanced Alert
- Order Entry + Cold State outreach (Experimental)
  Interventions: Other: Order Entry; Other: Cold State outreach; Other: Enhanced Alert
- Open Encounter + Cold State outreach (Experimental)
  Interventions: Other: Open Encounter; Other: Cold State outreach; Other: Enhanced Alert
- Order Entry + Simplified (Experimental)
  Interventions: Other: Order Entry; Other: Simplified; Other: Enhanced Alert
- Open Encounter + Simplified (Experimental)
  Interventions: Other: Open Encounter; Other: Simplified; Other: Enhanced Alert
- Order Entry + Sign-off alert (Experimental)
  Interventions: Other: Order Entry; Other: Sign-off alert; Other: Enhanced Alert
- Open Encounter + Sign-off alert (Experimental)
  Interventions: Other: Open Encounter; Other: Sign-off alert; Other: Enhanced Alert
- Order Entry + Pre-commitment (Experimental)
  Interventions: Other: Order Entry; Other: Pre-commitment; Other: Enhanced Alert
- Open Encounter + Pre-commitment (Experimental)
  Interventions: Other: Open Encounter; Other: Pre-commitment; Other: Enhanced Alert
- Order Entry + Different Risks (Experimental)
  Interventions: Other: Order Entry; Other: Different Risks; Other: Enhanced Alert
- Open Encounter + Different Risks (Experimental)
  Interventions: Other: Open Encounter; Other: Different Risks; Other: Enhanced Alert
- Standard Epic Basic Alert (Experimental)
  Interventions: Other: Order Entry; Other: Standard Epic Basic Alert
- No Alert (Usual Care) (No Intervention)

INTERVENTIONS:
Other: Order Entry — An alert will display in the electronic health record when the provider orders one of the high-risk medications for an eligible patient.
  Arms: Base Order Entry Alert; Order Entry + Cold State outreach; Order Entry + Different Risks; Order Entry + Follow-up booster Alert; Order Entry + Pre-commitment; Order Entry + Sign-off alert; Order Entry + Simplified; Standard Epic Basic Alert
Other: Open Encounter — An alert will display in the electronic health record when the provider opens the chart of an eligible patient.
  Arms: Base Open Encounter Alert; Open Encounter + Cold State outreach; Open Encounter + Different Risks; Open Encounter + Follow-up booster Alert; Open Encounter + Pre-commitment; Open Encounter + Sign-off alert; Open Encounter + Simplified
Other: Follow-up booster Alert — Once the order entry or open encounter alert displays, the provider will have the option to schedule a follow-up message that will be sent 4 weeks after the alert is triggered
  Arms: Open Encounter + Follow-up booster Alert; Order Entry + Follow-up booster Alert
Other: Cold State outreach — An in-basket message will be sent to the eligible provider 2 days before the eligible patient is scheduled for an in-person visit.
  Arms: Open Encounter + Cold State outreach; Order Entry + Cold State outreach
Other: Simplified — The alert language itself will be simplified.
  Arms: Open Encounter + Simplified; Order Entry + Simplified
Other: Sign-off alert — An alert will display in the electronic health record when the medication is sent to sign-off for providers.
  Arms: Open Encounter + Sign-off alert; Order Entry + Sign-off alert
Other: Pre-commitment — A two-staged pre-commitment electronic health record alert will be used. In the 1st alert, the providers will be prompted to discuss risks of these high-risk medications and share a handout about the risks with their patients, at their own discretion. The second alert will be either an order entry or open encounter alert, depending on the arm the provider is assigned to.
  Arms: Open Encounter + Pre-commitment; Order Entry + Pre-commitment
Other: Different Risks — Risks of the high-risk medications will be framed differently.
  Arms: Open Encounter + Different Risks; Order Entry + Different Risks
Other: Standard Epic Basic Alert — This alert will be representative of the alerts currently firing in the Atrius system and not incorporate any functionality.
  Arms: Standard Epic Basic Alert
Other: Enhanced Alert — An enhanced alert (known as a Best Practice Advisory [BPA]) will appear on the provider's electronic health record screen and will contain several standard components such as information about why the medication is dangerous for their patient and an order set that will allow providers to order a gradual dose taper for their patient, order alternative medications, place a referral to a behavioral health specialist, provide instructions on how to make lifestyle modifications to improve patient symptoms, and add patient instructions for how to gradually taper off benzodiazepines and sedative hypnotics, as applicable.
  Arms: Base Open Encounter Alert; Base Order Entry Alert; Open Encounter + Cold State outreach; Open Encounter + Different Risks; Open Encounter + Follow-up booster Alert; Open Encounter + Pre-commitment; Open Encounter + Sign-off alert; Open Encounter + Simplified; Order Entry + Cold State outreach; Order Entry + Different Risks; Order Entry + Follow-up booster Alert; Order Entry + Pre-commitment; Order Entry + Sign-off alert; Order Entry + Simplified

SUMMARY:
Prescribing of potentially unsafe medications for older adults is extremely common; benzodiazepines and sedative hypnotics are, for example, key drug classes frequently implicated in adverse health consequences for vulnerable older adults, such as confusion or sedation, leading to hospitalizations, falls, and fractures. Fortunately, most of these consequences are preventable. Physicians' lack of awareness of alternatives, ambiguous practice guidelines, and perceived pressure from patients or caregivers are among the reasons why these drugs are used more than might be optimal. Reducing inappropriate use of these drugs may be achieved through decision support tools for providers that are embedded in electronic health record (EHR) systems. While EHR strategies are widely used to support the informational needs of providers, these tools have demonstrated only modest effectiveness at improving prescribing. The effectiveness of these tools could be enhanced by leveraging principles of behavioral economics and related sciences.

DETAILED DESCRIPTION:
This is an adaptive cluster randomized control trial (RCT) to evaluate whether newly designed EHR-based tools designed using behavioral principles reduce inappropriate prescribing and adverse outcomes among older adults. This study will be conducted in outpatient and acute care practices of Atrius Health, a large integrated delivery network in eastern and central Massachusetts, which uses the Epic EHR system.

In Stage 1, approximately 200 primary care providers at Atrius Health will be randomized to receive usual care or an active intervention. Providers randomized to the active intervention will be randomly assigned to one of 15 active intervention arms. They will then be followed for 6 months. Providers randomized to one of the 15 active intervention arms will receive a newly-designed EHR tool to guide their care of eligible patients. Providers randomized to usual care will receive no newly-designed EHR tool. Providers will receive these EHR tools for their patients who meet the following criteria: 1) older adults (aged 65 years or more) and 2) who have been prescribed at least 90 pills of benzodiazepine or sedative hypnotic in the last 180 days.

At the end of Stage 1 follow-up, the 15 active intervention arms will be ranked based on their observed effectiveness at reducing prescribing high-risk medications and select up to the 5 more promising arms for Stage 2. In Stage 2, the providers assigned in Stage 1 to usual care will be randomized with equal probability to be assigned to one of the 5 most promising treatment arms identified or usual care. Providers randomized to one of up to the 5 selected treatment arms will receive an EHR tool to guide their care of eligible patients. After this analysis, the Stage 1 providers in the "winning" arms (i.e., the promising arms) will be randomly assigned to continue to receive their original treatment assignments or to usual care. Similarly, the Stage 1 providers assigned to treatment arms determined to be statistically inferior will be randomly assigned in equal proportions to one of the winning arms or to usual care.

After Stage 2, we will evaluate the effectiveness of the tools by comparing the effectiveness of the behavioral principles contained within the tools on outcomes, combining data across both Stages. This is our primary analytic approach.

No participant (patient or provider) provided consent for participation, as this trial received a waiver of informed consent and authorization for use of study data.

The Mass General Brigham trial described in the protocol is described in another clinicaltrials.gov record (NCT05538065).

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider at Atrius Health

Providers will receive these EHR tools for their patients who meet the following criteria:

1. older adults (aged 65 years or more)
2. who have been prescribed at least 90 pills of benzodiazepine or sedative hypnotic in the last 180 days.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atrius Health, Braintree, Massachusetts, United States

REFERENCES:
- [Derived] Lauffenburger JC, Isaac T, Trippa L, Glynn RJ, Russo M, Keller P, Robertson T, Kim DH, Bhatkhande G, Hanken KE, Haff N, Jungo KT, Crum KL, Blair MS, Brill G, Choudhry NK. Comparing Fourteen Behavioral Science Electronic Health Record Deprescribing Tools in Older Adults: NUDGE-EHR Adaptive Trial. J Am Geriatr Soc. 2025 Oct;73(10):3031-3043. doi: 10.1111/jgs.19609. Epub 2025 Jul 4. PMID 40614073
- [Derived] Lauffenburger JC, Isaac T, Trippa L, Keller P, Robertson T, Glynn RJ, Sequist TD, Kim DH, Fontanet CP, Castonguay EWB, Haff N, Barlev RA, Mahesri M, Gopalakrishnan C, Choudhry NK. Rationale and design of the Novel Uses of adaptive Designs to Guide provider Engagement in Electronic Health Records (NUDGE-EHR) pragmatic adaptive randomized trial: a trial protocol. Implement Sci. 2021 Jan 7;16(1):9. doi: 10.1186/s13012-020-01078-9. PMID 33413494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Atrius primary care providers were cluster-randomized to these arms based on data available from the electronic health record and were not recruited directly for the trial or evaluated for effectiveness outcomes. Patients were also not intervened upon nor directly enrolled into the study. As such, we received a waiver of informed consent for participation. The Mass General Brigham trial described in the protocol is a different record (NCT05538065).
Pre-assignment Details: Primary care providers were identified from electronic health record data and cluster randomized to a study arm in Stage 1. Patients who sought care from these primary care providers were identified based on electronic health record data for analyses. Providers were not assessed for effectiveness outcomes. After the interim analysis, primary care providers were re-randomized to a study arm in Stage 2.
Groups:
- No Alert (Usual Care): Providers randomized to usual care will receive no EHR tool, as is current clinical practice.
Period: Stage 1: October 2020-August 2021
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care)
Started (The numbers reflect the number of primary care providers assigned to each arm in Stage 1 of trial (n=201). Primary care providers were identified from electronic health record data and cluster randomized but were not evaluated for effectiveness outcomes. The number of patients cared for by these providers and evaluated for outcomes are shown in the next row ("Number of Patients Analyzed").) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 81
Number of Patients Analyzed (These are the number of patients analyzed for effectiveness outcomes from each arm of Stage 1. Patients were eligible for inclusion in the effectiveness evaluation if they met eligibility criteria based on electronic health record data, including being cared for by the providers in the row above. Patients were not directly intervened upon nor actively enrolled.) | 91 | 91 | 87 | 140 | 174 | 102 | 130 | 104 | 153 | 113 | 118 | 147 | 87 | 90 | 109 | 1173
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 81
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: September 2021-August 2022
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care)
Started (The numbers reflect the number of primary care providers assigned to each arm in Stage 2 of trial. As in Stage 1, providers were not evaluated for effectiveness outcomes. The number of patients cared for by them and evaluated for outcomes are shown in the next row. The number of providers in each arm for Stage 2 differs from Stage 1 because not all arms were selected for Stage 2, and not all of the providers from Stage 1 were eligible after interim analysis. 15 new providers were also added.) | 0 | 27 | 0 | 27 | 0 | 0 | 0 | 28 | 0 | 28 | 0 | 27 | 0 | 0 | 0 | 60
Number of Patients Analyzed (These are the number of patients analyzed for effectiveness outcomes from each arm of Stage 2. Patients were eligible for inclusion in the effectiveness evaluation if they met eligibility criteria based on electronic health record data, including being cared for by the providers in the row above. Patients were not directly intervened upon nor actively enrolled. These numbers represent unique patients not previously identified in Stage 1.) | 0 | 15 | 0 | 35 | 0 | 0 | 0 | 33 | 0 | 23 | 0 | 17 | 0 | 0 | 0 | 31
Completed | 0 | 27 | 0 | 27 | 0 | 0 | 0 | 28 | 0 | 28 | 0 | 27 | 0 | 0 | 0 | 60
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All of these baseline measures are for patients included in analyses across Stages 1 and 2 of the trial (n=3063 total, 2909 in Stage 1 and 154 in Stage 2). Data from primary care providers was not collected at baseline nor in follow-up. Baseline patient characteristics are shown for Stages 1 and 2 combined, as the analyses were pre-specified to be conducted combining outcomes across both Stages.
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care) | Total
Number analyzed (Participants) | 91 | 106 | 87 | 175 | 174 | 102 | 130 | 137 | 153 | 136 | 118 | 164 | 87 | 90 | 109 | 1204 | 3063
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (7.0) | 73.2 (6.3) | 73.7 (6.6) | 74.2 (6.8) | 74.4 (7.3) | 74.1 (7.4) | 7.7 (7.5) | 74.0 (7.1) | 75.5 (7.6) | 75.8 (7.7) | 72.9 (5.8) | 73.6 (7.1) | 75.6 (7.5) | 74.1 (7.5) | 77.0 (8.2) | 74.3 (7.0) | 74.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 73 | 53 | 129 | 145 | 56 | 87 | 110 | 101 | 100 | 80 | 106 | 58 | 44 | 73 | 759 | 2041
  Male | 24 | 33 | 34 | 46 | 29 | 46 | 43 | 27 | 52 | 36 | 38 | 58 | 29 | 46 | 36 | 445 | 1022
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian, Alaska Native, Native Hawaiian, or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 6
  Asian | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 23 | 45
  Black or African American | 2 | 2 | 5 | 4 | 5 | 7 | 4 | 2 | 2 | 4 | 1 | 7 | 3 | 2 | 3 | 31 | 84
  White | 86 | 93 | 69 | 163 | 144 | 87 | 118 | 126 | 147 | 123 | 112 | 149 | 80 | 82 | 93 | 1051 | 2723
  More than one race | 1 | 3 | 2 | 1 | 4 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 5 | 24 | 47
  Unknown or Not Reported | 0 | 5 | 5 | 5 | 18 | 2 | 4 | 5 | 0 | 5 | 3 | 2 | 1 | 3 | 1 | 50 | 109
  Hispanic | 1 | 2 | 4 | 0 | 1 | 2 | 3 | 1 | 0 | 4 | 2 | 3 | 2 | 0 | 3 | 21 | 49
Benzodiazepine quantity: Number of pills prescribed in past 180 days measured in EHR system [Mean (Standard Deviation); unit: number of pills prescribed] | 187.9 (135.9) | 200.0 (118.6) | 186.9 (116.4) | 195.6 (118.2) | 222.0 (293.3) | 218.0 (233.2) | 209.9 (175.4) | 199.2 (122.6) | 214.5 (158.0) | 185.1 (115.7) | 227.7 (151.2) | 205.2 (145.5) | 220.3 (155.4) | 229.7 (220.0) | 190.5 (119.9) | 203.1 (149.4) | 205.2 (162.0)
Sedative hypnotic quantity: Number of pills prescribed in past 180 days measured in EHR system [Mean (Standard Deviation); unit: number of pills prescribed] | 132.1 (70.9) | 154.4 (71.3) | 143.4 (66.6) | 138.0 (64.3) | 153.3 (87.7) | 107.5 (31.5) | 130.0 (74.1) | 150.1 (76.5) | 145.0 (53.6) | 154.9 (81.9) | 172.7 (73.2) | 136.8 (55.3) | 146.8 (64.7) | 150.7 (64.9) | 162.3 (100.7) | 147.6 (73.7) | 147.1 (72.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Inappropriate Prescribing by Study Arm: Descriptive Comparison Across Study Arms
Description: This outcome is measured as a composite of 1) discontinuation of study high-risk medications (i.e., active discontinuation or lack of an order during follow-up) or 2) ordering a dose taper (for benzodiazepine or sedative hypnotics) using EHR data by the primary care provider included in the study arm. If any of these actions occurred by the primary care provider, then the patient was considered to have had a change in prescribing (i.e., a reduction in inappropriate prescribing). This outcome was measured as a binary outcome. As noted in the Outcome Measure Time Frame below, these outcomes were measured and presented across both stages of the adaptive trial at Atrius Health rather than separately, as this was part of the pre-specified analytic plan.
Time Frame: 22 months (2 stages)
Population: Patients who met eligibility criteria for inclusion in the analysis (adults ≥65 years, who were prescribed ≥90 pills of benzodiazepine or sedative hypnotic in the last 180 days and had an office or telemedicine visit with a primary care provider who was assigned to a study arm), as measured from EHR system data across Stages 1 and 2
Measure: Number; unit: percentage of patients
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care)
Number analyzed (Participants) | 91 | 106 | 87 | 175 | 174 | 102 | 130 | 137 | 153 | 136 | 118 | 164 | 87 | 90 | 109 | 1204
percentage of patients | 35.2 | 33 | 35.6 | 40.6 | 25.9 | 39.2 | 42.3 | 38 | 27.5 | 29.4 | 33.9 | 45.1 | 28.7 | 32.2 | 30.3 | 33.6

2. Primary Outcome: Change in Inappropriate Prescribing by the Seven Behavioral Intervention Factors (Open Encounter Timing, Boostering, Cold-state Priming, Simplification, Sign-off Approval, Pre-commitment, and Risk Framing): Primary Analysis Approach
Description: This outcome is measured as a binary composite of 1) discontinuation of study high-risk medications (i.e., active discontinuation or lack of an order during follow-up) or 2) ordering a dose taper using EHR data by the primary care provider in the arm. If the provider performed any of these actions, then the patient was considered as having a change in prescribing (i.e., a reduction in inappropriate prescribing). As noted in the Time Frame below, these outcomes were measured and analyzed across both Stages of the trial in the primary analysis. The following outcomes are shown stratified by patients who were in arms containing one of the seven behavioral intervention factors and also among those in arms that did not contain an intervention factor. The primary analysis conducts analyses by intervention factor; the model treats patients in arms that do not contain any of the behavioral factors (i.e., Base Order Entry Alert, Standard Epic Basic Alert, and Usual Care) as the referent.
Time Frame: 22 months (2 stages)
Population: Patients who met eligibility criteria for inclusion in the analyses (adults ≥65 years, who were prescribed ≥90 pills of benzodiazepine or sedative hypnotic in the last 180 days and had an office or telemedicine visit with a primary care provider in the trial), as measured in the EHR across Stages 1 and 2. These groups are not mutually exclusive as the study arms could contain multiple intervention factors (e.g., Open Encounter Timing and Boostering); thus, the overall total exceeds 3063.
Measure: Number; unit: percentage of patients
Groups:
- Timing (Open Encounter): Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including timing (at encounter opening vs. ordering a medication as the referent). The number of participants reported here represents the number of patients whose primary care providers received an Open Encounter alert. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed.
- Boostering: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including boostering (i.e., receiving a follow-up message) vs. not having boostering as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert that contained boostering. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed.
- Cold-state Priming: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including cold-state priming (i.e., receiving a message in advance) vs. not having cost-state priming as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert containing cold-state priming. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed.
- Simplification: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including simplification (i.e., having simplified language included in the alert) vs. not having simplification as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert containing simplification. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed.
- Sign-off Approval: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including sign-off approval (i.e., having an additional alert with sign-off approval) vs. not having sign-off approval as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert containing sign-off approval. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed.
- Pre-commitment: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including precommitment (i.e., receiving an alert first requesting a patient discussion followed by a subsequent deprescribing action) vs. not having precommitment as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert containing precommitment. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed
- Risk Framing: Each study arm was categorized based on whether it included one of seven different behavioral science components (or "intervention factors"), including risk framing (i.e., receiving an alert with an alternative risk presentation) vs. not having risk framing as the referent. The number of participants reported here represents the number of patients whose primary care providers received an alert containing alternative risk framing. Note that some individual alerts contained multiple behavioral intervention factors (i.e., intervention factors are not mutually exclusive); therefore, the number of participants reported in this table sum to be greater than the number of total patient participants analyzed
- No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care): The numbers reported here reflect the participants in the Base Order Entry Alert, Standard Epic Basic Alert, and Usual Care arms, which did not have any of the behavioral intervention factors. Analyses were conducted based on individual behavioral intervention factors, not at the study arm level. Thus, the effect of each intervention factor was evaluated relative to patients in those arms that did not contain those intervention factors. This included patients in the Base Order Entry Alert, Standard Epic Basic Alert, and Usual Care arms as well as any arm that did not have that intervention factor.
Arm/Group | Timing (Open Encounter) | Boostering | Cold-state Priming | Simplification | Sign-off Approval | Pre-commitment | Risk Framing | No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care)
Number analyzed (Participants) | 910 | 262 | 276 | 267 | 289 | 282 | 177 | 1404
percentage of patients | 33.1 | 38.9 | 30.8 | 40.1 | 28.4 | 40.4 | 30.5 | 33.5
Statistical Analysis 1: Comparison: Timing (Open Encounter) vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); Outcomes were evaluated using generalized linear mixed models with a logit link and binary errors, evaluating the association between the intervention factors (i.e., behavioral components) and the primary outcome, pooling across both stages of the trial and adjusting for provider-level clustering; Test type: Superiority; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.97 to 1.49] — The Odds Ratio compares having "open encounter" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having an "open encounter" alert in the arm they were assigned to
Statistical Analysis 2: Comparison: Boostering vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); Outcomes were evaluated using generalized linear mixed models with a logit link and binary errors, evaluating the association between the intervention factors (i.e., behavioral components) and the primary outcome, pooling across both stages of the 2-stage Atrius adaptive trial and adjusting for provider-level clustering. As noted in our Study Protocol and pre-specified, the analyses are conducted across the intervention factors across the study arms, rather than between the study arms; Test type: Superiority; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.83 to 1.59] — The OR compares between having "boostering" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "boostering" in the arm they were assigned to
Statistical Analysis 3: Comparison: Cold-state Priming vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.61 to 1.16] — The OR compares between having "cold-state priming" as an intervention factor in the arm the patient's primary care providers were assigned to vs. all others not having "cold-state priming" in the arm they were assigned to
Statistical Analysis 4: Comparison: Simplification vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.88 to 1.64] — The OR compares between having "simplification" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "simplification" in the arm they were assigned to
Statistical Analysis 5: Comparison: Sign-off Approval vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.52 to 0.98] — The OR compares between having "sign-off approval" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "sign-off approval" in the arm they were assigned to
Statistical Analysis 6: Comparison: Pre-commitment vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.89 to 1.64] — The OR compares between having "pre-commitment" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "pre-commitment" in the arm they were assigned to
Statistical Analysis 7: Comparison: Risk Framing vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 2, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.55 to 1.19] — The OR compares patients having "risk framing" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "risk framing" in the arm they were assigned to

3. Secondary Outcome: Quantity of Prescribing by Study Arm: Descriptive Comparison Across Study Arms
Description: This outcome is measured on the patient level as the number of cumulative lorazepam milligram equivalents of high-risk medications prescribed to patients by Atrius providers over the follow-up for the relevant adaptive trial stage, measured within the EHR system. This outcome was measured as a continuous outcome. As noted in the Outcome Measure Time Frame below, these outcomes were measured and presented across both stages of the adaptive trial at Atrius Health rather than separately, as this was part of the pre-specified analytic plan.
Time Frame: 22 months (2 stages)
Population: Among eligible study population included (adults ≥65 years, who were prescribed ≥90 pills of benzodiazepine or sedative hypnotic in the last 180 days and had an office or telemedicine visit with a primary care provider assigned to that study arm), as measured from the EHR system across Stages 1 and 2 of the trial.
Measure: Mean (Standard Deviation); unit: Cumulative lorazepam mg equivalents
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care)
Number analyzed (Participants) | 91 | 106 | 87 | 175 | 174 | 102 | 130 | 137 | 153 | 136 | 118 | 164 | 87 | 90 | 109 | 1204
Cumulative lorazepam mg equivalents | 64.5 (87.6) | 119.8 (179.7) | 94.4 (176.5) | 104.7 (170.0) | 156.6 (207.5) | 146.3 (425.3) | 114.2 (181.6) | 110.0 (160.3) | 114.6 (188.7) | 93.6 (147.0) | 107.0 (180.8) | 121.1 (196.7) | 82.0 (90.2) | 118.0 (166.5) | 123.6 (214.4) | 114.4 (194.9)

4. Secondary Outcome: Quantity of Prescribing by the Seven Behavioral Intervention Factors (Open Encounter Timing, Boostering, Cold-state Priming, Simplification, Sign-off Approval, Pre-commitment, and Risk Framing): Primary Analysis Approach
Description: This outcome is measured on the patient level as the cumulative number of lorazepam milligram equivalents of high-risk medications prescribed to patients by Atrius providers over the follow-up for the relevant adaptive trial stage, measured in the EHR system. This outcome was measured as a continuous outcome. As noted in the Time Frame below, these outcomes were measured and analyzed across both Stages of the trial in the primary analysis. The following outcomes are shown stratified by patients who were in arms containing one of the seven behavioral intervention factors and also among those in arms that did not contain an intervention factor. The primary analysis conducts analyses by intervention factor; the model treats patients in arms that do not contain any of the behavioral factors (i.e., Base Order Entry Alert, Standard Epic Basic Alert, and Usual Care) as the referent.
Time Frame: 22 months (2 stages)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cumulative lorazepam mg equivalents
Arm/Group | Timing (Open Encounter) | Boostering | Cold-state Priming | Simplification | Sign-off Approval | Pre-commitment | Risk Framing | No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care)
Number analyzed (Participants) | 910 | 262 | 276 | 267 | 289 | 282 | 177 | 1404
Cumulative lorazepam mg equivalents | 114.5 (215.1) | 101.3 (171.9) | 152.8 (305.9) | 112.0 (170.7) | 104.7 (170.4) | 115.2 (190.0) | 100.3 (135.4) | 111.9 (191.8)
Statistical Analysis 1: Comparison: Timing (Open Encounter) vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); Outcomes were evaluated using generalized linear mixed models with an identity link and normally-distributed errors, evaluating the association between the intervention factors (i.e., behavioral components) and secondary outcome, pooling across both stages of the 2-stage Atrius adaptive trial and adjusting for provider-level clustering. As noted in our Study Protocol and pre-specified, the analyses are conducted across intervention factors across study arms, rather than between the study arms; Test type: Superiority; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-17.6 to 21.2] — The estimate compares having "open encounter" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "open encounter" in the arm they were assigned to
Statistical Analysis 2: Comparison: Boostering vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-41.8 to 17.5] — The estimate compares having "boostering" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "boostering" in the arm they were assigned to
Statistical Analysis 3: Comparison: Cold-state Priming vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 39.5, 95% CI 2-sided [11.6 to 67.4] — The estimate compares having "cold-state priming" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "cold-state priming" in the arm they were assigned to
Statistical Analysis 4: Comparison: Simplification vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-30.4 to 26.9] — The estimate compares having "simplification" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "simplification" in the arm they were assigned to
Statistical Analysis 5: Comparison: Sign-off Approval vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-37.6 to 17.4] — The estimate compares having "sign-off approval" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "sign-off approval" in the arm they were assigned to
Statistical Analysis 6: Comparison: Pre-commitment vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-24.1 to 32.5] — The estimate compares having "pre-commitment" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "pre-commitment" in the arm they were assigned to
Statistical Analysis 7: Comparison: Risk Framing vs No Behavioral Factor (Base Order Entry Alert, Standard Epic Basic Alert, Usual Care); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -12.0, 95% CI 2-sided [-45.5 to 21.5] — The estimate compares having "risk framing" as an intervention factor in the arm the patients' primary care providers were assigned to vs. all others not having "risk framing" in the arm they were assigned to

ADVERSE EVENTS:
Time Frame: 22 months (2 stages) - these outcomes were measured across both stages of the 2-stage Atrius adaptive trial. The Mass General Brigham trial described in the Study Protocol is listed under a different clinicaltrials.gov record (NCT05538065), as that is a distinct trial.
Description: Deaths and adverse events are reported for patients who were included in the analyses for the trial. Deaths and adverse events were not collected, monitored, or assessed for providers. For patients, we used an automatic adverse event reporting system to monitor for any AEs that occurred, which were routinely reviewed by quality and safety specialists at the institution. In addition, for patients, we retrospectively identified patient deaths through a retrospective review within the EHR.
Arm/Group | Base Order Entry Alert | Base Open Encounter Alert | Order Entry + Follow-up Booster Alert | Open Encounter + Follow-up Booster Alert | Order Entry + Cold State Outreach | Open Encounter + Cold State Outreach | Order Entry + Simplified | Open Encounter + Simplified | Order Entry + Sign-off Alert | Open Encounter + Sign-off Alert | Order Entry + Pre-commitment | Open Encounter + Pre-commitment | Order Entry + Different Risks | Open Encounter + Different Risks | Standard Epic Basic Alert | No Alert (Usual Care)
All-Cause Mortality (participants affected / at risk) | 1/91 | 2/106 | 1/87 | 2/175 | 0/174 | 1/102 | 4/130 | 5/137 | 1/153 | 11/136 | 2/118 | 6/164 | 0/87 | 0/90 | 2/109 | 18/1204
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/106 | 0/87 | 0/175 | 0/174 | 0/102 | 0/130 | 0/137 | 0/153 | 0/136 | 0/118 | 1/164 | 0/87 | 0/90 | 0/109 | 0/1204
Other Adverse Events (participants affected / at risk) | 0/91 | 0/106 | 0/87 | 0/175 | 0/174 | 0/102 | 0/130 | 0/137 | 0/153 | 0/136 | 0/118 | 0/164 | 0/87 | 0/90 | 0/109 | 0/1204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Base Order Entry Alert (N=91) | Base Open Encounter Alert (N=106) | Order Entry + Follow-up Booster Alert (N=87) | Open Encounter + Follow-up Booster Alert (N=175) | Order Entry + Cold State Outreach (N=174) | Open Encounter + Cold State Outreach (N=102) | Order Entry + Simplified (N=130) | Open Encounter + Simplified (N=137) | Order Entry + Sign-off Alert (N=153) | Open Encounter + Sign-off Alert (N=136) | Order Entry + Pre-commitment (N=118) | Open Encounter + Pre-commitment (N=164) | Order Entry + Different Risks (N=87) | Open Encounter + Different Risks (N=90) | Standard Epic Basic Alert (N=109) | No Alert (Usual Care) (N=1204)
Intentional overdose (Psychiatric disorders) | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | 1 | NA | NA | NA | NA — Intentional overdose of several prescription medications, including benzodiazepine. Deemed unrelated to the intervention by the DSMB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04284553/Prot_SAP_000.pdf